CLINICAL TRIAL: NCT00352482
Title: Sildenafil Treatment in Patients With Idiopathic Pulmonary Fibrosis and Pulmonary Hypertension - a Pilot Cross-over Study
Brief Title: Sildenafil to Increase Exercise Capacity in Individuals With Idiopathic Pulmonary Fibrosis and Pulmonary Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 414; P50HL067665-05 (NIH)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2007-12

CONDITIONS: Pulmonary Fibrosis; Hypertension, Pulmonary
Keywords: Pulmonary Hypertension; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Hypertension, Pulmonary; Idiopathic Pulmonary Fibrosis | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil (50 mg)

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic lung disease that affects an individual's ability to breathe. Currently, no medications can reverse the damage to the lungs caused by IPF, but individuals are encouraged to engage in moderate exercise to strengthen lung function. This study will evaluate the effectiveness of sildenafil at improving exercise tolerance and breathing difficulties in individuals with IPF.

DETAILED DESCRIPTION:
IPF is a disease that damages the air sacs in the lungs and leads to widespread and permanent scarring of lung tissue. Individuals with IPF may experience breathing difficulties, cough, chest pain, and a decreased exercise capacity. There is no cure for this disease, and individuals usually die within 3 to 5 years. It is recommended that individuals with IPF engage in moderate exercise, as this can help maintain strength and improve lung function. Many individuals with IPF also suffer from pulmonary hypertension, which is high blood pressure in the arteries leading to the lungs. Sildenafil, a medication currently used to treat pulmonary hypertension, increases blood flow to the lungs and enhances gas exchange within the lungs. The purpose of this study is to evaluate the effectiveness of sildenafil at improving exercise tolerance and breathing difficulties in individuals with IPF and pulmonary hypertension.

This 3-week study will enroll individuals with IPF and pulmonary hypertension. Study visits will occur at baseline, and Weeks 1 and 2. At the baseline visit, participants will perform a 6-minute walk test, which will measure the distance walked in a 6-minute period. Oxygen levels will be measured prior to and during the test, and standardized questionnaires will be completed to assess breathing difficulties. A second 6-minute walk test will be performed 1 hour following the first test. At the Week 1 visit, participants will be randomly assigned to receive a single dose of either 50 mg of sildenafil or placebo. One hour after receiving the medication, they will complete another 6-minute walk test. The Week 2 visit will be identical to the Week 1 visit, except participants who received sildenafil at Week 1 will receive placebo at Week 2, and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* IPF, diagnosed according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) consensus statement (with or without surgical lung biopsy)
* Pulmonary hypertension, defined as mean pulmonary artery pressure (MPAP) greater than or equal to 25 mm Hg by right heart catheterization (RHC)

Exclusion Criteria:

* Interstitial lung disease due to conditions other than IPF
* Recent lung or upper respiratory tract infection within 4 weeks of study entry
* Acute or chronic impairment other than dyspnea (e.g., angina pectoris, intermittent claudication) limiting the ability to comply with study requirements (e.g., 6-minute walk test)
* Known hypersensitivity to sildenafil
* Known or suspected coronary artery disease (CAD)
* Unstable angina
* Nitrate use
* Known or suspected aortic stenosis (AS)
* Known or suspected heart attack, stroke, or life-threatening arrythmias within 1 month of study entry
* Severe chronic heart failure, defined as New York Heart Association (NYHA) class III/IV and/or left ventricular ejection fraction less than 25%
* Known penile deformities
* Known kidney or liver dysfunction
* Uncontrolled diabetes (blood glucose less than 60 mg/dl or greater than 300 mg/dl)
* Severe serum sodium abnormalities (serum sodium less than 130 mEq/L or greater than 150 mEq/L)
* Condition that may predispose participant to priapism (e.g., sickle cell anemia, multiple myeloma, leukemia)
* Retinitis pigmentosa
* Known or suspected idiopathic hypertrophic subaortic stenosis (IHSS)
* Low blood pressure (systolic blood pressure [SBP] less than 100 mm Hg or diastolic blood pressure [DBP] less than 50 mm Hg)
* Uncontrolled systemic high blood pressure (SBP greater than 180 mm Hg or DBP greater than 100 mm Hg)
* Cardiopulmonary rehabilitation program started within 8 weeks of study entry or likely to start prior to the conclusion of the study
* Treatment with an endothelin receptor antagonist, iloprost, epoprostenol, inhibitors of CYP3A4 (e.g., cimetidine, erythromycin, ketoconazole, itraconazole, mibefradil), protease inhibitors (e.g., amprenavir, indinavir, or ritonavir), rifampin, alpha-blockers (e.g., doxazosin), or other phosphodiesterase-5 inhibitors
* Current use of alcohol, grapefruit juice, or St. John's wort
* Pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (measured at Week 3)

SECONDARY OUTCOMES:
Oxygen saturation (SpO2) at rest
Lowest SpO2 with exertion (measured during 6-minute walk test)
Total duration of SpO2 below 89% with exertion (measured during 6-minute walk test)
Recovery time (measured during 6-minute walk test)
Mean SpO2 and area under the curve (measured during 6-minute walk test)
Desaturation index (measured by the 6-minute walk distance multiplied by the SpO2 mean value)
Level of breathlessness (measured by Borg dyspnea index questionnaire) (all measured at Week 3)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Zisman, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pulmonary Outpatient Clinic,, Los Angeles, California, United States

REFERENCES:
- [Derived] Collard HR, Anstrom KJ, Schwarz MI, Zisman DA. Sildenafil improves walk distance in idiopathic pulmonary fibrosis. Chest. 2007 Mar;131(3):897-899. doi: 10.1378/chest.06-2101. PMID 17356110
- See also: Click here for the Coalition for Pulmonary Fibrosis web site — http://www.coalitionforpf.org